CLINICAL TRIAL: NCT02060851
Title: Effects of Early Parenteral Iron Combined Erythropoietin in Preterm Infants
Brief Title: Effects of Early Short-term Intravenous Iron Supplements Combined EPO in Preterm Infants
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kunshan First People's Hospital Affiliated to Jiangsu University (Industry)
Responsible Party: Principal Investigator, Wang Hua, Ethics Committee of Kunshan First People's Hospital, Kunshan First People's Hospital Affiliated to Jiangsu University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: kunshan002
Record Dates: First submitted 2014-02-09; First posted 2014-02-12 (Estimated); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Malnutrition
Keywords: EPO; Intravenous iron; iron storage; preterm anemia
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Vifor and EPO (Experimental): intravenous iron and EPO
  Interventions: Drug: Vifor and EPO
- control (Placebo Comparator): no intravenous iron or EPO
  Interventions: Other: standard PN
- Vifor (Experimental): intravenous iton but no EPO
  Interventions: Drug: Vifor

INTERVENTIONS:
Other: standard PN — Group 1: a control group who received standard PN
  Other Names: a control group
  Arms: control
Drug: Vifor — iron sucrose, 200 μg/kg per day, was given everyday with PN,
  Other Names: an iron-supplemented group
  Arms: Vifor
Drug: Vifor and EPO — EPO, 400U/kg, was given twice a week (Monday and Friday). IS, 200 μg/kg per day, was given everyday with PN, and the dose was continued until 2 weeks after birth
  Other Names: iron-supplemented combined EPO group
  Arms: Vifor and EPO

SUMMARY:
There are wide variations in iron supplementation practices in NICU.Guidelines on pediatric Parenteral nutrition suggested the dose of 200μg/kg.d iron by parenteral nutrition.

DETAILED DESCRIPTION:
The study was approved by the ethics committee of Xinhua Hospital, and all parents gave written informed consent.

Study Design This was a randomized, controlled, double-blind, interventional trial of iron (iron sucrose) supplementation given from age of 1 day until full 2 weeks to preterm infants in NICU, who divided into three groups, control(PN without iron and EPO), Vifor and vifor and EPOE group, according to the recommended dosage of ESPEN .

Outcome Measures General information and indicators including anemia iron storage were measured. And the same time oxidative stress indicators were monitored at age of 1day and 2 weeks.

General growth parameters including the blood sugar, liver and renal function index before and after the intervention were tested.

Hematological evaluation including RBC, Hb, MCV, MCH, MCHC, RET, CRP were mesured before and after the intervention. The three groups were all peripheral blood.

Iron storage evaluation including ferritin, serum iron, TIBC on the days were measured before and after the intervention. We used the radio-immunoassay method to test the ferritin (DADE BEHRING, Germany), the chemical method to the serum iron and the automatic biochemical analyzer (automatic biochemical analyzer, 7600, HITACH).

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants with birth weight less than 2.5kg Have parenteral nutrition indication With written informed consent of parents or guardian

Exclusion Criteria:

* Kidney and liver function abnormal have hemolytic disease have hemorrhagic disease have Serious congenital malformation have septicemia have plethora newborn use TPN less than ten days

Max Age: 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 96 (Actual)
Dates: Start 2014-02; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Number of participants with Hematological evaluation | up to 2 weeks
  Hematological evaluation including RBC, Hb, MCV, MCH, MCHC, RET, CRP were measured before and after the intervention. The three groups were all peripheral blood.

SECONDARY OUTCOMES:
Iron storage | up to 2 weeks
  Iron storage evaluation including ferritin, serum iron, TIBC on the days were measured before and after the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Kunshan First Hospital, Kunshan, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No